CLINICAL TRIAL: NCT06357520
Title: An Open-label, Fixed Sequence Study in Healthy Participants to Assess the Pharmacokinetics of Baxdrostat When Administered Alone and in Combination With Itraconazole
Brief Title: A Study to Investigate the Pharmacokinetics of Baxdrostat When Given Alone and in Combination With Itraconazole in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D6970C00005
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baxdrostat and Itraconazole (Experimental): Participants will receive single dose of baxdrostat tablet orally on Day 1 in Period 1, followed by itraconazole capsule orally twice a day on Day 6 and once daily on Days 7 to 8 in Period 2, and then single dose of baxdrostat tablet orally on Day 9 with itraconazole capsule orally once daily on Days 9 to 16 in Period 3.
  Interventions: Drug: Baxdrostat; Drug: Itraconazole

INTERVENTIONS:
Drug: Baxdrostat — Baxdrostat tablet will be administered orally.
  Other Names: CIN-107
Drug: Itraconazole — Itraconazole capsule will be administered orally.

SUMMARY:
The main purpose of this study is to assess the effect of itraconazole on the pharmacokinetic (PK) of baxdrostat.

DETAILED DESCRIPTION:
This study will be an open-label, 3-period fixed sequence study conducted at a single Clinical Unit.

The study will comprise of:

* A Screening Period of maximum 28 days
* Period 1: Period 1 will start from Day -1 to Day 6 (followed by pharmacokinetic (PK) sampling of baxdrostat). Baxdrostat administration on Day 1 to Day 6
* Period 2: Period 2 will start from Day 6 (after the last PK sample in period 1) to Day 8. Itraconazole administration on Days 6 to 8 (twice a day [BID] on Day 6 and once daily [QD] on Days 7 and 8)
* Period 3: Period 3 will start from Day 9 to Day 17. Baxdrostat administration on Day 9 and itraconazole administration on Days 9 to 16 QD
* A Final Follow-up Visit at 7 to 14 days after the last baxdrostat PK sample in Period 3

All participants will receive 2 single doses of baxdrostat and 12 doses of itraconazole, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female participants of non-childbearing potential aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* All female participants must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit (Study Day -1).
* Have a body mass index between 18 and 32 kilograms per meter square (kg/m2) inclusive and weigh greater than or equal to (>=) 50 kilograms (kg) and less than or equal to <=) 120 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the principal investigator (PI), may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of drug-related hepatic toxicity.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* History of any treatment with QT prolongation drugs.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to baxdrostat or itraconazole.
* Participants who have previously received baxdrostat.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Area Under Plasma Concentration-Time Curve From Time Zero To Infinity (AUCinf) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The effect of itraconazole on the PK (AUCinf) of baxdrostat will be assessed.
Maximum Observed Plasma Drug Concentration (Cmax) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The effect of itraconazole on the PK (Cmax) of baxdrostat will be assessed.

SECONDARY OUTCOMES:
Extrapolated Area Under The Curve From Tlast to Infinity (AUCextr) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (AUCextr) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Area Under Plasma Concentration Curve from Time Zero to the Last Quantifiable Concentration (AUClast) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (AUClast) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Apparent Total Body Clearance (CL/F) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (CL/F) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Apparent Volume Of Distribution Based On The Terminal Phase (Vz/F) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (Vz/F) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Terminal Elimination Half-life (t1/2λz) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (t1/2λz) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Terminal Rate Constant (λz) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (λz) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Mean Residence Time (MRTinf) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (MRTinf) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Time To Reach Maximum Observed Concentration (tmax) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (tmax) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Ratio of Baxdrostat (Baxdrostat + Itraconazole) to Baxdrostat (Alone) Based on Maximum Plasma Concentration (RCmax) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (RCmax) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Ratio of Baxdrostat (Baxdrostat + Itraconazole) to Baxdrostat (Alone) Based on AUClast (RAUClast) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (RAUClast) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Ratio of Baxdrostat (Baxdrostat + Itraconazole) to Baxdrostat (Alone) Based on AUCinf (RAUCinf) | Period 1: Days 1 to 6 (pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, and 120 hours post-dose); Period 3: Days 9 to 17 (pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 hours)
  The PK (RAUCinf) of baxdrostat when baxdrostat is administered alone or in combination with itraconazole will be evaluated.
Number of Participants with Adverse Events | Up to 8 weeks
  The safety and tolerability of baxdrostat alone and in combination with itraconazole will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/